CLINICAL TRIAL: NCT05135598
Title: Partners For Life: Off-line Health Promotion Program for Ultra-orthodox Jewish Women During the COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Donna R Zwas (Other)
Responsible Party: Sponsor-Investigator, Donna R Zwas, Principle Investigator, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020123-HMO-CTIL
Record Dates: First submitted 2021-09-02; First posted 2021-11-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Pre-post evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health behavior change intervention (Experimental): Participants will receive a pedometer, workbook, partner, and 15 weekly phone group meetings.
  Interventions: Other: Partners for Life health behavior change program

INTERVENTIONS:
Other: Partners for Life health behavior change program — A health behavior change intervention based on partner learning, utilizing low-tech media and a workbook.

SUMMARY:
The purpose of this study is to evaluate a unique culturally-tailored intervention aimed at increasing healthy eating and physical activity in Ultra-Orthodox Jewish women during the COVID-19 pandemic. Utilizing a pre-post study design, this intervention is based on the CDC's Diabetes Prevention Program (DPP) and integrates low-tech media, partner learning, group support, and practical workbook content.

DETAILED DESCRIPTION:
UOJ women in Israel have poorer health outcomes and sub-optimal health behaviors than their counterparts. Contributing factors to these disparities include poverty, limited access to information, and insufficient culturally-appropriate opportunities. COVID-19 has exacerbated this inequity, with reduced income, opportunities and time availability, as well as increased weight, social isolation, loss, stress and emotional issues. While COVID-19 brought these health issues to the forefront, they are ongoing - and currently overlooked.

The purpose of this study is to evaluate a unique culturally-tailored intervention aimed at increasing healthy eating and physical activity in Ultra-Orthodox Jewish women during the COVID-19 pandemic. Utilizing a pre-post study design, this intervention is based on the CDC's Diabetes Prevention Program (DPP) and integrates low-tech media, partner learning, group support, and practical workbook content. Participants are recruited through an Ultra-orthodox Jewish continuing education institution for women and either register with a friend or are assigned a partner. Each woman receives a pedometer and workbook with information and skill-building worksheets to complete weekly in pairs (via phone or in person). All dyads will join weekly phone-based group meetings led by a group leader, to share challenges and successes as well as problem solve. It is hypothesized that this intervention will increase the targeted health behaviors as well as reduce weight in participants.

ELIGIBILITY:
Inclusion Criteria: Females aged 18-85, willingness to commit to participation in the lifestyle intervention and follow-up.

-

Exclusion Criteria: Pregnancy, history of schizophrenia, severe depression, untreated bipolar disorder, end-stage renal disease, type 1 diabetes, unstable angina, congestive heart failure, inability to participate in the group without assistance, dementia, inability to communicate in Hebrew.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who self-represent as female will be eligible.
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Healthy Heart Score | At intervention completion after 15 weeks
  The Healthy Heart Score is a lifestyle-based CVD prediction model that was developed using health data from 61,025 women in the Nurses' Health Study and 34,478 men in the Health Professionals Follow-up Study, who were free of chronic disease in 1986 and followed for CVD for up to 24 years. The Healthy Heart Score is based on the diet and lifestyle factors that include smoking, weight, exercise, and intake of alcohol, fruits and vegetables, whole grains, nuts, sugary beverages, and red and processed meat. On a prospective study, women with higher predicted CVD risk based on the Healthy Heart Score had an 18-fold higher risk of type 2 diabetes mellitus,5-fold higher risk of hypertension, and 3-fold higher risk of hypercholesterolemia during 20 years.
Eating Behavior | At intervention completion after 15 weeks
  The Dutch Eating Behavior Questionnaire (DEBQ) is a measure of Restrained, External, and Emotional eating. This questionnaire has good internal consistency and factorial validity as well as predictive validity for food consumption.
Pedometer Steps | At intervention completion after 15 weeks
  Pedometer steps (measured with the Omron pedometer Model HJ-320) will provide an objective measure of increased physical activity. Omron pedometers have been shown to demonstrate validity and reliability at various mounting positions in both healthy and overweight adults. Participants in all groups will be reminded to wear the pedometer for the week before each data collection point to assess average weekly step count. Intervention participants will also provide weekly step count data throughout the intervention. Measures will include average daily steps, as an objective measure of physical activity, and percentage change in steps, as an objective measure of change in physical activity level.
Energy Expenditure | At intervention completion after 15 weeks
  The Ministry of Health (as well as the World Health Organization) recommends engaging in at least 150 minutes of moderate physical activity or 75 minutes of vigorous physical activity per week. Exercising at the level of 500 MET-minutes per week has been defined as the threshold for an average reduction of 20% to 30% in mortality risk and exercise may have comparatively increased benefits in women compared to men. Energy expenditure will be assessed by the self-administered Women's Health Initiative Physical Activity Questions (WHI-PAQ), measuring recreational physical activities. The Women's Health Initiative was a pivotal, prospective study of women's health, including the impact of health behavior on cardiovascular health54. The WHI PAQ has been validated compared to accelerometry and has been shown to be reliable. Metabolic equivalents (METs) will be calculated based on energy expenditure related to these activities using standardized classifications.

SECONDARY OUTCOMES:
Emotion Regulation Skills | At intervention completion after 15 weeks
  The Difficulties in Emotion Regulation Scale-16 (DERS-16) is a brief measure of emotion regulation difficulties. This scale demonstrates good internal consistency, test-retest reliability, as well as convergent and discriminant validity.
Body Mass Index (BMI) | At intervention completion after 15 weeks
  Weight will be measured in kilograms using a standardized, calibrated scale and height will be measured using a standardized stadiometer. Weight loss in kilograms and percent weight loss will be calculated. BMI will be calculated by body weight /height2, and change in BMI will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD, Principal Investigator — Hadassah
Locations (1):
- Hadassah University Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neamah HH, Sebert Kuhlmann AK, Tabak RG. Effectiveness of Program Modification Strategies of the Diabetes Prevention Program: A Systematic Review. Diabetes Educ. 2016 Apr;42(2):153-65. doi: 10.1177/0145721716630386. Epub 2016 Feb 15. PMID 26879459
- [Background] Chiuve SE, Cook NR, Shay CM, Rexrode KM, Albert CM, Manson JE, Willett WC, Rimm EB. Lifestyle-based prediction model for the prevention of CVD: the Healthy Heart Score. J Am Heart Assoc. 2014 Nov 14;3(6):e000954. doi: 10.1161/JAHA.114.000954. PMID 25398889